CLINICAL TRIAL: NCT06959134
Title: Community Health Workers-led Multicomponent Intervention for Hypertension Control in Rwanda: A Cluster Randomized Controlled Trial.
Brief Title: Community Health Workers-led Multicomponent Intervention for Hypertension Control in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rwanda (Other)
Responsible Party: Principal Investigator, MWISENEZA Innocent, PhD Student, Rwanda Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 695/CMHS IRB/2024
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Community Health Workers; Multicomponent Intervention; Hypertension; Randomized clinical trials; Control
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An experimental arm will be composed with 100 patients with uncontrolled blood pressure (Experimental): In the intervention arm patients with uncontrolled hypertension will be getting routine care form the NCD clinic at the health center and in addition to this , they will receive an assistance from the community health workers where they will give the patients health education mainly on lifestyle modifications, medication adherence and self monitoring of blood pressure at home for detecting the variability and report them accordingly.
  Interventions: Behavioral: The intervention will be mainly focused on the lifestyle modification and medication adherence, and self monitoring at home
- In this arm which will be no intervention, there will be100 patients with uncontrolled hypertension (No Intervention): In this arm patient will receive the routine care from the health center NCD clinic and at the end of the study data collection period , data will be compared to those blood pressure measurement from the intervention group

INTERVENTIONS:
Behavioral: The intervention will be mainly focused on the lifestyle modification and medication adherence, and self monitoring at home — In the intervention arm, study participants will received health education mainly based on lifemodification changes which will include; eating healthy diet, adopting healthy physical exercise, smoking cessation , moderate alcohol consumption and stress amanagement), and will be taugh on medication adherence, but also on self monitoring of blood pressure for detecting the variation and react accordingly.
  Arms: An experimental arm will be composed with 100 patients with uncontrolled blood pressure

SUMMARY:
This study will involve patients, families and healthcare providers in the following ways

1. Patients; The main study participants will be patients with uncontrolled hypertension who are currently managed at the health center level. After being enrolled in the study the patients will be asked to follow the recommendations given by healthcare providers and community health workers during the study period(Intervention group follow up of one year), and will be required to continuously respect the standard appointment at the health center and in addition to this they will be visited by community health workers at their household at least once per month, and during this visit they will have a health education basically on medication adherence and lifestyle modifications including adopting a culture of healthy physical activity for better control of hypertension not only this but community health worker will take one measurement on Blood pressure in between the month in addition to the usual measurement taken at the health center at the time of the regular appointment. And then on this side everytime the community health worker will visit a patient , family member will be requested to be present for helping to remind the patient the healthy habit discussed as most of these patients are old requiring a close follow up.
2. Family; Will play a key role in helping the patient to adopt new healthy habit depending on the preference and reminding the patient on adhering to medications regimen but also notify the community health worker or the research if there is any adverse health outcome occured during the research period.
3. Health care provider; This will involves healthcare providers on different level mainly the Community health workers and Nurses working in Non Communicable disease Clinic at the health centers.

Methods: A cluster randomized controlled trial will be randomly assigned to four health centers in the intervention arm and another four health centers for routine health care hypertensive care, enrolling 25 patients with uncontrolled hypertension per health center, equivalent to 200 total sample size.

Participants: Patients with uncontrolled hypertension followed-up from health centers non-communicable disease (NCD) clinics in eight health centers(Gihogwe, Kagugu, Remera and Bumbogo in Gasabo and Nyamata, Mayange, Gashora and Ntarama health center in Bugesera district.

Interventions: Participants in the intervention arm will receive an integrated community health worker led- multicomponent intervention (CHW led-MCI) which includes CHW-led home-based intervention including health coaching, monthly home blood pressure monitoring and feedback, lifestyle changes and medication adherence. While those in the control arm received routine health center nurse led management of hypertension in Non-communicable diseases (NCD) clinics ('standard of care').

Outcomes: Effectiveness of the CHW led-MCI will be evaluated through three main research objectives and their outcomes. To evaluate if Integrated CHW led-MCI can control hypertension will be measured through primary outcome clinical outcomes are (i) the difference in the proportion of patients with controlled hypertension (< 130/80 mmHg) between the CHW led-MCI intervention and control groups at 3, 6, 9 and 12 months and secondary on lowing blood pressure, mean blood pressure will be reported, dietary sodium consumption, glucose, BMI as well as improving medication adherence between the CHW led-MCI intervention and control groups at 3, 6, 9 and 12 months (Objective 1). We will explore the facilitators and barriers in the implementation of CHW-led MCI to control hypertension at Rwandan health centers from the patient, health center nurses, facility managers, and policymakers perspectives (objective 2). Finally, we will evaluate the cost, effectiveness, and cost-effectiveness of CHW-led MCI implementation outcomes to inform policymakers on a scale out of the intervention (objective 3).

Study utility: This study will help policymakers to understand if the recent task-shifting of nurses to manage hypertension at the health center level is working as well as generate additional evidence on CHW-led intervention to improve hypertension control at the community/household level in Rwanda and other low-resource countries.

DETAILED DESCRIPTION:
This randomised controlled trials will be conducted in eight health centers, and will have three main sub studies:

The first substudy will mainly evaluate the community health workers multicomponent intervention, which will assist the routine care patients receive from the health centers provided by nurses to control hypertension, especially those patients with uncontrolled hypertension. These will include home visits, health education, monitoring blood pressure at home and physical activity of these patients.

Substudy two; this substudy will mainly consist of the evaluation of facilitators and barriers which may be implicated in the community health workers multicomponent intervention to control hypertension among hypertensive patients. This part will be a qualitative study where the investigator will evaluate the opinion of patients , NCD clinic nurses at health centers, health center managers but also policymakers perspectives in the ministry of health about the multicomponent intervention. And each group of participants will mention the possible facilitators and barriers which may make this intervention to run smoothly and therefore benefit patients.

Sub study three; This part will evaluate the financial burden means that A health system perspective system will be used to determine the cost, effectiveness, and cost-effectiveness of CHW-led multicomponent intervention on uncontrolled hypertensive patients attending Rwanda health centers. Participants' data will be used to estimate CHWs-led MCI effects and HTN control. It's main objective will be to determine the cost, effectiveness, and cost-effectiveness of CHW-led multicomponent intervention on hypertensive patients attending Rwanda health centers

ELIGIBILITY:
Inclusion Criteria:

* Blood Pressure above or equal to 130/80
* Male and female aged 21 years old and above
* Patients attending NCD clinics in the eight selected Rwanda health centers during the period of data collection.

Exclusion Criteria:

* Blood Pressure below 130/80 mmHg
* Patients without other adult living in the same house
* Hypertensive patients with active systemic illness (fever, known liver disease), clinically unstable heart failure, advanced CKD
* Patients deemed mentally unfit.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with controlled hypertension and mean blood pressure between intervention and control group | This will be measured at 3 , 6 and 12 months from the time of data collection
  the difference in the proportion of patients with controlled hypertension (< 130/80 mmHg) between the CHW led-MCI intervention and control groups at 3, 6, 9 and 12 months and secondary on lowing blood pressure, mean blood pressure will be reported, BMI as well as improving medication adherence between the CHW led-MCI intervention and control groups at 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Facilitators and barriers in the implementation of community health workers-led multicomponents intervention to control hypertension among uncontrolled hypertensive patients | Data will be collected from the 3 to 6 months of data collection
  We will explore the facilitators and barriers in the implementation of CHW-led MCI to control hypertension at Rwandan health centers from the patient, health center nurses, facility managers, and policymakers perspectives.
  The outcome will be measured using an interview guide to conduct interview and FGD. Interview guides (IDIs and FGDs will be developed in accordance with previous literature reviews and research on CHW-led MCI).The PI will collect the data, assisted by a trained research assistant. All interviews will held in a nearby, quiet, and convenient room for the study participants. All interviews will be audio-recorded and transcribed verbatim in Kinyarwanda (the local language) to English. However, the work will be re-evaluated again by the PI and double-checked by the research supervisors. The transcripts will be loaded into the NVivo 11 software for coding and data analysis.We will use these coding to find connections between themes and identify overarching principles.

OTHER OUTCOMES:
Cost, effectiveness and cost effectiveness of community health workers led multi components intervention | Will be evaluated retrospectively for the past 12 months following data collection from the intervention and control group
  QALYs will be the primary measurement of efficacy outcomes. The incremental cost-effectiveness ratio (ICER) between the multicomponent intervention and normal care will be computed by dividing the cost difference by the difference in efficacy in quality-adjusted life years (QALYs). One-way sensitivity analysis will be used to address methodological and individual parameter uncertainties. A tornado diagram analysis will be conducted to determine the relative weight of each variable in terms of total uncertainty. Parameters for sensitivity analyses will be chosen based on systematic fluctuations around the basic model's parameters or disparities between trial data and published studies. The parameters investigated by one-way sensitivity analysis will include time horizon, discount rate for costs and QALYs, transition probabilities, relative risk of HTN events, and HTN. When 95% confidence intervals are available, they will be used to calculate ranges for 1-way sensitivity analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Richard KALISA, PhD, Study Director — University of Rwanda/School of Public Health; Clarisse Marie Claudine SIMBI, PhD, Study Director — University of Rwanda/School of Public Health; Kevin NWANNA, PhD, Study Director — University of Rwanda/ School of Public Health
Locations (1):
- Gasabo and Bugesera health centers, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No
To ensure the privacy of study participants, the individual participant data will not be shared but also as one of the requirements of the clinicalTrials.gov